CLINICAL TRIAL: NCT06193473
Title: Evaluation Of Clinical Pharmacy Services in Patients Receiving Antithrombotic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Muhammed Yunus BEKTAY, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pharm. Role in Cardiology
Record Dates: First submitted 2023-12-05; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases; Drug Use
Keywords: clinical pharmacist; antithrombotic drugs; drug-related problems; cardiovascular diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Group in which only observation is made by the clinical pharmacist (No Intervention): For patients in this group, no intervention (i.e. recommendation) will be made to physicians by the clinical pharmacist. Within the intervention group, patient characteristics such as the length of hospital stay, reason for hospitalization, underlying conditions, and the appropriateness of prescribed medications were evaluated for the patients who received antithrombotic treatment and met the inclusion criteria. The participant will take standard treatment. Evaluations will be recorded. Follow-up was performed to determine whether the patients had a re-admission within 3 months.
- Intervention Group: Group to which the clinical pharmacist makes recommendations (Experimental): For patients in this group, intervention (i.e. recommendation) will be made to physicians by the clinical pharmacist. Within the intervention group, patient characteristics such as the length of hospital stay, reason for hospitalization, underlying conditions, and the appropriateness of prescribed medications were evaluated for the patients who received antithrombotic treatment and met the inclusion criteria. Through medication reviews, evaluations were made to identify drug-related problems and provide solutions to these problems. The clinical pharmacist provided recommendations to the physicians regarding significant clinically important problems. Additionally, follow-up was performed to determine whether the patients had a re-admission within 3 months.
  Interventions: Behavioral: Intervention Group: Group to which the clinical pharmacist makes recommendations

INTERVENTIONS:
Behavioral: Intervention Group: Group to which the clinical pharmacist makes recommendations — The drugs administered to patients within 24-48 hours after hospitalization were recorded. A detailed medication review will be conducted by the clinical pharmacist during the participants' hospitalization.As a result of a comprehensive evaluation, recommendations were made to doctors regarding drug-related problems and were recorded.
  Arms: Intervention Group: Group to which the clinical pharmacist makes recommendations

SUMMARY:
Clinical pharmacy services aim to enhance patient outcomes and reduce the risk of potential drug-related harm by offering patient-centred pharmaceutical care. In the hospital setting, clinical pharmacists collaborate with physicians as part of a multidisciplinary team to identify and prevent DRPs (Drug-related problems). Clinical pharmacist interventions encompass 'any action initiated by a pharmacist that directly results in patient management or a modification in medication.' The favourable clinical and economic impacts of interventions have been well-established for decades. Clinical pharmacists have played an important role in ensuring the effective and correct use of medicines in many settings.

This study aims to investigate the clinical pharmacy services provided by clinical pharmacists to patients receiving antithrombotic therapy. For this study, patients were divided into two groups: a control group and an intervention group. A comprehensive medication review will be conducted by the clinical pharmacist for both the control and intervention groups. Drug-related problems such as drug selection, dose errors, possible drug-drug interactions, and inappropriate drug use, will be identified. In the control group, no interventions will be made by the clinical pharmacist. In the intervention group, solution recommendations for identified and clinically significant issues will be presented to the physician, and the provided services will be documented. Furthermore, the groups will be evaluated for whether there are any hospital readmissions within 1 and 3 months following discharge for the patients.

DETAILED DESCRIPTION:
Patients with cardiovascular disease are at significant risk for adverse drug events and medication errors. Moreover, the rate of use of high-risk drugs such as antithrombotic drugs is higher in these patients. In the literature, antithrombotics have been shown as one of the main causes of adverse drug events and drug-related hospitalizations. Therefore, follow-up of patients treated with antithrombotics is very important. Guideline-based therapy significantly reduces the risk of all-cause and cardiovascular (CV) death. Multidisciplinary antithrombotic management can play an important role in increasing prescribing physicians' adherence to guidelines. Effective interventions such as medication review, establishment of treatment protocols, education, and medication reconciliation at hospitalization and discharge can help increase adherence to the guideline. In patients receiving antithrombotic therapy, individual evaluation of drug therapy suitability, formulation of a drug treatment plan, dose adjustment, drug monitoring, detection and prevention of clinically important drug-drug interactions, and antithrombotic transition protocols should be considered. Such interventions must appropriately balance each individual's risk of thromboss and bleeding.

Pharmacists are recognized as leading healthcare professionals in detecting, resolving, and preventing DRPs. Assessments of the quality and value of pharmacist interventions remain crucial for the development of new pharmaceutical care services and for enhancing our understanding of the frequency and variety of DRPs observed in various clinical settings. The literature has demonstrated the impact of Clinical Pharmacy Services on cardiovascular patients. Collaborating with a clinical pharmacist during inpatient treatment has been shown to improve medication adherence, reduce adverse drug reactions, and minimize medication errors post-discharge. The benefits of these pharmacist-led services in reducing hospitalization and healthcare costs were emphasized. Clinical pharmacy services have contributed to an enhancement in healthcare quality without compromising patient well-being. Pharmacists can take on the responsibility of antithrombotic management, ensuring that patients receive the right medication, in the correct dosage, and for the appropriate duration from the initial consultation to outpatient follow-up. Increasing the continuity of pharmaceutical care will enhance patient outcomes and reduce costs.

In this study, two groups were established as control group and intervention group. In the control group, no interventions will be made by the Clinical Pharmacist. Within the intervention group, patient characteristics such as the length of hospital stay, reason for hospitalization, underlying conditions, and the appropriateness of prescribed medications were evaluated for the patients who received antithrombotic treatment and met the inclusion criteria. Through medication reviews, evaluations were made to identify drug-related problems and provide solutions to these problems. The clinical pharmacist provided recommendations to the physicians regarding significant clinically important problems. Additionally, follow-up was performed to determine whether the patients had a re-admission within 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years and older.
* Receiving antithrombotic treatment.
* Having complete biochemical and complete blood count values collected at least twice, with two-day medication information fully entered into the hospital system.
* Patients who could be evaluated by the clinical pharmacist for at least 24 hours within the intervention group.

Exclusion Criteria:

* Being under 18 years old.
* Not using antithrombotic medication.
* Patients whose biochemical and complete blood count values were not collected twice and whose two-day medication information was not fully recorded in the hospital system.
* Patients in the intervention group whom the clinical pharmacist did not see for at least 24 hours (weekend hospital admission followed by Monday morning discharge, Friday admission with weekend discharge, etc.) were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Acceptance rate of suggested intervention (number) | From the date of randomization until there are 200 patient participants in each group. Average 1 year.
  Acceptance rate of suggested intervention. Medication-related problems and recommendations are classified according to PCNE (Pharmaceutical Care Network Europe) version 9.1. It was recorded how many suggestions were made in the intervention group and how many of these suggestions were accepted.
Length of hospital stay (days) | From date of randomization until the date of discharge from the hospital, assessed up to 1 year.
  Length of hospital stay
Within three months readmission (number of patients re-admitted to hospital) | Whether patients were readmitted to the hospital within three months of discharge or transfer.
  In order to determine which group of patients has the highest number of hospital re-admissions and to evaluate whether there is a significant difference between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Fikret Vehbi Izzettin, Prof.Dr., Principal Investigator — Bezmialem Vakıf Üniversitesi
Locations (1):
- Bezmialem Vakıf Üniversitesi, Istanbul, Fatih, Turkey (Türkiye)